CLINICAL TRIAL: NCT07066072
Title: The Radiofrequency Therapy in Management of Sickle Cell Disease Chronic Pain
Brief Title: The Radiofrequency Therapy in Management of Sickle Cell Disease Chronic Pain RCT Tested the Effect of TECAR Therapy on Sickle Cell Disease Chronic Pain.
Acronym: RCT/TECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mai mohamed abdelhamed, assisstant lecturer mai mohamed abdelhamed pediatric department principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC No: MD-45-2023; REC No: MD-45-2023 (Registry Identifier: cairo university)
Record Dates: First submitted 2025-04-18; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: the Use of Radiofrequency Ablation in Form of TECAR(Capacitive and Resistive Transfer Energy) in Chronic Pain of Sickle Cell Disease Patients
Keywords: radiofrequency; sickle cell disease; chronic pain
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): the control group will have no intervention will be on standard of care therapy known for sickle cell disease meaning pharmacological therapy in form of hydroxyurea,analgesics and blood transfusion.
  Interventions: Other: standard pharmacological therapy in sickle cell disease like hydroxyurea,paracetamol,ibubrofen and blood transfusion if needed
- TECAR group (Active Comparator): the tecar group will receive 12 sessions of Tecar therapy (TECAR: Capacitive and Resistive Energy Transfer) over totally 6 weeks (2 sessions/week)
  Interventions: Device: Tecar therapy (TECAR: Capacitive and Resistive Energy Transfer).

INTERVENTIONS:
Device: Tecar therapy (TECAR: Capacitive and Resistive Energy Transfer). — the Tecar therapy (TECAR: Capacitive and Resistive Energy Transfer) will be assigned to TECAR group
  Arms: TECAR group
Other: standard pharmacological therapy in sickle cell disease like hydroxyurea,paracetamol,ibubrofen and blood transfusion if needed — this is the standard medical care assigned to control group
  Arms: control group

SUMMARY:
The goal of this clinical trial study is to assess effect of radiofrequency on chronic pain of sickle cell disease pain .

All SCA participants who fulfilled inclusion and exclusion criteria were 220; only 170 participant agreed to consent for the study .

Participants who seek frequent medical attention were included in the TECAR group without randomization and they were 15 patients, and the rest of the participants (155 patient) were randomized according to the following ratio as 1:1.2 respectively for both arms arm1: the TECAR group arm 2: the control group .

The main questions to answer are:

primary outcome measure: assess short term effect of TECAR therapy on chronic sickle cell diaease chronic pain by assessment of change in pain scores following 1st TECAR session.

secondary outcomes: assess long term effect of TECAR therapy by assessment of change in chronic pain scores along overall period of study (6weeks).

TECAR (Capacitive and Resistive Energy Transfer device) used:

(C-200 Capenergy Spain)

participants: 2 arms : one arm: TECAR group. 2nd arm: control group. one arm: received TECAR therapy in addition to the standard of care for SCA (hydroxyurea, analgesics [NSAIDs or paracetamol], and blood transfusion on demand).

The second arm received standard of care only. tools used to assess pain:

1. VAS questionnaire.
2. BPI questionnaire.
3. HRQOL questionnaire.

DETAILED DESCRIPTION:
This randomized non blinded controlled study was conducted as collaboration between Haematology department in Cairo university Children hospital and the Anaesthesia department in Cairo university hospital from the period between 2022&2024 patients were recruited from Haematology clinic who fulfilled inclusion criteria in absence of exclusion criteria.

Inclusion criteria:

1. All types of sickle cell disease (SS/SB0/SB+/SS trait)
2. Age of participants ranging from 6 years to 30 years.
3. SCA participants with known and unknown cause of chronic pain

Exclusion criteria:

1. Those participants with associated chronic disease or end organ damage.
2. participants in acute Vaso occlusive crisis.
3. Participants on antiepileptics or antidepressant drugs.

Participants and grouping:

This study investigated the effect of Transcutaneous Electrical Capacitive Resistive (TECAR) therapy on chronic pain in 170 Sickle Cell Anemia (SCA) participants.

TECAR session:

These sessions were done for TECAR group participants on a fixed site of pain which was back and lower limbs. The participants were lying in a supine position, and the session is done for around 40 minutes in 2 positions consequently (each site 20 minutes).

Drainage position: The capacitive plates were inserted over the sole of feet while the passive plate was inserted under the back facing lumbar vertebrae for 20 minutes. The temperature was adjusted to 37OC.

The frequency selected was one of three available frequencies (0.8, 1, or 1.2 megahertz) associated with the highest tissue uptake (the frequency associated with the greatest number of light arrows on the right screen of each channel).

Low back position: the capacitive and resistive probes were placed blindly over the most tender areas and temperature was adjusted to 41OC for 20 minutes.

Immediately before and 30 minutes after each session VAS was recorded for pain assessment.

ELIGIBILITY:
Inclusion Criteria:

1. All types of sickle cell disease (SS/SB0/SB+/SS trait)
2. Age of patients ranging from 6 years to 30 years.
3. SCA patients with known and unknown cause of chronic pain

Exclusion Criteria:

1. Those patients with associated chronic disease or end organ damage.
2. patients in acute Vaso occlusive crisis.
3. Patients on antiepileptics or antidepressant drugs.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
primary outcome was defined as successful treatment, indicated by patients exhibiting a VAS score below 4 at 30 minutes following the initial first TECAR therapy session. | 30 minutes
  We categorized the patients studied according to change in the recorded VAS score between before 1st session and 30 minutes after the first session into the following five subgroups:
  1. st group: VAS turned to 0.
  2. nd group: VAS turned out to be less than 4.
  3. rd group: VAS turned to 4.
  4. th group: VAS turned to above 4.
  5. th group: VAS remained the same.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt